CLINICAL TRIAL: NCT01159171
Title: Phase II Study of the Combination of Bevacizumab (rhuMab VEGF) and Oxaliplatin Plus Capecitabine (XELOX) in Patients With Advanced Colorectal Cancer
Brief Title: A Study of Avastin (Bevacizumab) and Oxaliplatin Plus Xeloda (Capecitabine) in Patients With Advanced Colorectal Cancer.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18523
Record Dates: First submitted 2010-07-07; First posted 2010-07-09 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Capecitabine; Oxaliplatin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]; Drug: capecitabine [Xeloda]; Drug: oxaliplatin

INTERVENTIONS:
Drug: bevacizumab [Avastin] — 5 mg/kg intravenously every 14 days
Drug: capecitabine [Xeloda] — 1000 mg/m2 orally b.i.d. , Days 1 - 14 of every 28-day cycle
Drug: oxaliplatin — 40 mg/m2 iv weekly

SUMMARY:
This study will assess the efficacy and safety of treatment with the combination Avastin (bevacizumab) 5mg/kg iv every 2 weeks, Xeloda (capecitabine) 1000 mg po b.i.d. on Days 1-14 of every 28-day cycle and oxaliplatin 40mg/m2 iv weekly in patients with inoperable locally advanced or metastatic colorectal cancer. The anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >=18 years of age
* Locally advanced or metastatic colorectal cancer
* No previous treatment with chemotherapy for metastatic disease
* Measurable and/or evaluable lesions

Exclusion Criteria:

* Radiotherapy within 4 weeks before study
* Untreated brain metastases or primary brain tumors
* Chronic, daily treatment with high-dose aspirin (>325mg/day)
* Co-existing malignancies, or malignancies diagnosed within the last 5 years, with the exception of basal and squamous cell cancer, or cervical cancer in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Italy (6):
  - Aviano
  - Fano
  - Palermo
  - Rimini
  - Roma
  - Torino

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Oxaliplatin + Capecitabine: Participants received bevacizumab 5 milligrams per kilograms (mg/kg) intravenously (IV) on Days 1 and 15; oxaliplatin 40 mg per square meter (mg/m^2) IV on Days 1, 8, 15, and 22; and capecitabine 1000 mg/m^2 orally (PO) twice daily (BID) on Days 1 through 14 followed by 2 weeks without treatment. This cycle was repeated until disease progression, unacceptable toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Started | 50
Completed | 0
Not Completed | 50
Not completed — Adverse Event | 11
Not completed — Progression of Disease | 28
Not completed — Protocol Violation | 1
Not completed — Need for Surgery | 5
Not completed — Medical Decision | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least one dose of one study medication.
Groups:
- Bevacizumab + Oxaliplatin + Capecitabine: Participants received bevacizumab 5 mg/kg IV on Days 1 and 15; oxaliplatin 40 mg/m^2 IV on Days 1, 8, 15, and 22; and capecitabine 1000 mg/m^2 PO BID on Days 1 through 14 followed by 2 weeks without treatment. This cycle was repeated until disease progression, unacceptable toxicity, or participant withdrawal.
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.08 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR was defined as the percentage of participants who achieved complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). CR was defined as disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR was defined as greater than or equal to (≥)30 percent (%) decrease under baseline of the sum of the longest diameter (LD) diameters of all target lesions. No unequivocal progression of non-target disease. No new lesions. Complete and partial responses must have been confirmed no less than 4 weeks after the criteria for response were first met.
Time Frame: Baseline, every 3 months to progression of disease or end of study (up to 24 months)
Population: Intent to Treat (ITT) Population: all participants who signed the informed consent, were assigned a study patient number, and who were administered at least 1 dose of 1 study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
percentage of participants | 42.86 [0.31 to NA]
Statistical Analysis 1: Comparison: Bevacizumab + Oxaliplatin + Capecitabine; Test type: Superiority or Other; p = 0.0047, One sample exact binomial test — One-sided p-value

2. Secondary Outcome: Duration of Response - Percentage of Participants With an Event by 24 Months
Description: Duration of overall response (CR or PR) was calculated only for participants of the ITT population whose best overall response was CR or PR based on RECIST criteria. Duration of overall response was defined as the time from the date of the first assessment of CR or PR status until the date of progression or death. Data for participants who were alive without any objectively documented disease progression at the end of the study were censored as of the date of last contact.
Time Frame: Baseline, every 3 months to progression of disease or end of study (up to 24 months)
Population: ITT population; only participants with a best overall response of CR or PR were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 21
percentage of participants | 57.14

3. Secondary Outcome: Duration of Response
Description: Duration of overall response (CR or PR) was calculated for participants of the ITT population whose best overall response was CR or PR based on RECIST criteria. Duration of overall response was defined as the time from the date of the first assessment of CR or PR status until the date of progression or death. Data for participants who were alive without any objectively documented disease progression at the end of the study were censored as of the date of last contact. Mean time to event was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 3 months to progression of disease or end of study (up to 24 months)
Population: ITT Population; only participants with a best overall response of CR or PR were included in the analysis.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 21
months | 8.31 (1.97)

4. Secondary Outcome: Duration of Stable Disease - Percentage of Participants With an Event by 24 Months
Description: Duration of stable response (CR, PR, or stable disease [SD]) was calculated only for participants of the ITT population whose best overall response was CR, PR, or SD based on RECIST criteria. Duration of overall response was defined as the time from the date of the first assessment of CR, PR, or SD status until the date of progression or death. Data for participants who were alive without any objectively documented disease progression at the end of the study were censored as of the date of last contact.
Time Frame: Baseline, every 3 months to progression of disease or end of study (up to 24 months)
Population: ITT Population; only participants with a best overall response of CR, PR, or SD were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 40
percentage of participants | 52.50

5. Primary Outcome: Percentage of Participants by Best Overall Response
Description: Best response recorded from the start of treatment until disease progression. Based on assessment of CR, PR, stable disease (SD), or progressive disease (PD), according to RECIST. CR: disappearance of all target lesions, non-target lesions, and normalization of tumor marker level. PR: ≥30% decrease under baseline of the sum of the LD diameters of all target lesions. CR and PR persist on repeat imaging study at least 4 weeks after initial documentation. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. Reference is the smallest sum LD. PD: at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum longest diameter recorded or the appearance of one or more new lesions.
Time Frame: Baseline, every 3 months to progression of disease or end of study (up to 24 months)
Population: ITT Population. 5 participants were not assessed as they did not reach the 3 month time-point.
Measure: Number; unit: percentage of participants
Groups:
- Bevacizumab + Oxaliplatin + Capecitabine: Cycle 1 (28-Day Cycle) Participants received 5 milligrams/kilograms (mg/kg) bevacizumab intravenously (IV) on Days 1 and 15; 40 mg/meter^2 (mg/m^2) oxaliplatin IV on Days 1, 8, 15, and 22; and 2000 mg/m^2 capecitabine orally (PO) in a divided dose every 12 hours within 30 minutes following a meal, on Days 1 through 14 followed by a rest period on Days 15 through 28. Cycle 1 was repeated until disease progression, unacceptable toxicity, or participant withdrawal.
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
percentage of participants
  CR | 4.08
  PR | 38.78
  SD | 38.78
  PD | 8.16

6. Secondary Outcome: Duration of Stable Disease
Description: Duration of stable response (CR, PR, or SD) was calculated only for participants of the ITT population whose best overall response was CR, PR, or SD based on RECIST criteria. Duration of overall response was defined as the time from the date of the first assessment of CR, PR, or SD status until the date of progression or death. Data for participants who were alive without any objectively documented disease progression at the end of the study were censored as of the date of last contact. Mean time to event was estimated using the Kaplan-Meier method.
Time Frame: Baseline, every 3 months to progression of disease or end of study (up to 24 months)
Population: ITT Population: only participants with a best overall response of CR, PR, or SD were included in the analysis.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 40
months | 10.09 (1.30)

7. Secondary Outcome: Time to Treatment Failure (TTF) - Percentage of Participants With an Event by 24 Months
Description: TTF was defined as the time in months from Day 1 until discontinuation of treatment for any reasons. These reasons included: death due to any cause, treatment toxicity (adverse event), insufficient therapeutic response (progression of disease), failure to return (lost to follow-up), refusing treatment (participant non-compliance), being unwilling to cooperate and withdrawing consent (participant withdrew consent).
Time Frame: Baseline, every month to end of treatment (up to 24 months)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
percentage of participants | 81.63

8. Secondary Outcome: Time to Treatment Failure
Description: TTF was defined as the time in months from Day 1 until discontinuation of treatment for any reasons. These reasons included: death due to any cause, treatment toxicity (adverse event), insufficient therapeutic response (progression of disease), failure to return (lost to follow-up), refusing treatment (participant non-compliance), being unwilling to cooperate and withdrawing consent (participant withdrew consent). Mean TTF was estimated using the Kaplan-Meier method.
Time Frame: Baseline, monthly to end of study (up to 24 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
months | 7.44 (0.84)

9. Secondary Outcome: Time to Progression (TTP) - Percentage of Participants With an Event by 24 Months
Description: TTP was defined as the time time in months from Day 1 until the date of first documented progressive disease, or death due to any cause. Data for participants who were alive without disease progression at the end of study, or who were non-responder participants (without tumor assessment after baseline) were censored at Day 1.
Time Frame: Baseline, monthly to end of study (up to 24 months)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
percentage of participants | 91.84

10. Secondary Outcome: Time to Progression
Description: TTP was defined as the time in months from Day 1 until the date of first documented progressive disease, or death due to any cause. Data for participants who were alive without disease progression at the end of study, or who were non-responder participants (without tumor assessment after baseline) were censored at Day 1. Mean TTP was estimated using the Kaplan-Meier method.
Time Frame: Baseline, monthly to end of study (up to 24 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
months | 9.61 (0.90)

11. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event by 24 Months
Description: OS was defined as the time in months from Day 1 until the date of death due to any cause. Data for participants who were alive at the end of the study were censored at the date of the last available follow-up visit.
Time Frame: Baseline, monthly to end of study (up to 24 months)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
percentage of participants | 89.90

12. Secondary Outcome: Overall Survival
Description: OS was defined as the time in months from Day 1 until the date of death due to any cause. Data for participants who were alive at the end of the study were censored at the date of the last available follow-up visit. Mean OS was estimated using the Kaplan-Meier method.
Time Frame: Baseline, monthly to end of study (up to 24 months)
Population: ITT Population
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Number analyzed (Participants) | 49
months | 20.23 (1.68)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected form the date of first study-drug intake until 28 days after the date of last study-drug intake.
Description: All participants who received at least 1 dose of study treatment were included in the safety population. Nonserious AEs presented in this record include all AEs reported during the study, not just nonserious events.
Arm/Group | Bevacizumab + Oxaliplatin + Capecitabine
Serious Adverse Events (participants affected / at risk) | 18/49
Other Adverse Events (participants affected / at risk) | 48/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Oxaliplatin + Capecitabine (N=49)
Angina pectoris (Cardiac disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 3
Pain (General disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Oxaliplatin + Capecitabine (N=49)
Anaemia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 14
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 22
Gingival bleeding (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 19
Stomatitis (Gastrointestinal disorders) | 5
Subileus (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 15
Asthenia (General disorders) | 11
Fatigue (General disorders) | 9
Mucosal inflammation (General disorders) | 9
Pyrexia (General disorders) | 12
Influenza (Infections and infestations) | 4
Blood alkaline phosphatase increased (Investigations) | 4
Blood lactate dehydrogenase increased (Investigations) | 4
Neutrophil count (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 4
Neuropathy peripheral (Nervous system disorders) | 13
Paraesthesia (Nervous system disorders) | 22
Sciatica (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 12
Phlebitis (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.